CLINICAL TRIAL: NCT03875586
Title: EMOCONSULT : Consultation Reasons in Family Medicine, a Tunisian National Survey
Brief Title: Consultation Reasons in Family Medicine
Acronym: EMOCONSULT
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Tunisian Society of Family Medicine (STMF) (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-005-EMOCONSULT
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Evaluate the Reasons for Consultation in Family Medicine
Keywords: Reasons for consultation; Family Medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Tunisian society of family medicine STMF proposes to coordinate a national, observational, transversal and multicenter survey, at the consultations of general medicine / family medicine.

DETAILED DESCRIPTION:
The Tunisian society of family medicine STMF proposes to coordinate a national, observational, transversal and multicenter survey carried out during two weeks, at the consultations of general medicine / family medicine. The main objective of the survey is to describe the reasons for consultation in general medicine / family medicine. The results obtained from this survey will make it possible to specify the specificities inherent to the reasons for consultations of Tunisians but especially to the peculiarities of the local health system (public and private). This survey will help us to assimilate our practices and harmonize them in order to optimize patient care and reposition family medicine in the patient's care path as well as the degree of adherence of practitioners to international recommendations in the care of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed consent, read and signed

Exclusion Criteria:

• Consent not obtained

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients consulting in general medicine / family medicine.
Sampling Method: Non-Probability Sample
Enrollment: 10822 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Describe the reasons for consultation in family medicine / general medicine | 2 weeks
  All patients presenting in consultation in general medicine / family medicine will be recruited in the survey in order to describe the different reasons for consultation

CONTACTS AND LOCATIONS:
Overall Officials: Maha Ben Moallem Hachicha, MD, Study Chair — STMF; Zied Ben Lamine, MD, Study Chair — STMF
Locations (2):
- Tunisia (2):
  - STMF - Société Tunisienne de Médecine de Famille, Tunis
  - DACIMA, Tunis

REFERENCES:
- See also: STMF FB page — https://www.facebook.com/STMF.TN/